CLINICAL TRIAL: NCT04464746
Title: Therapeutic Adherence in Uncontrolled Arterial Hypertension: Selective Detection by Urine Antihypertensive Drugs or Metabolits Analysis and Effectiveness of a Program to Improve Compliance
Brief Title: Therapeutic Adherence in Uncontrolled Arterial Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Fondo de Investigacion Sanitaria (Other)
Responsible Party: Principal Investigator, Anna Oliveras, Head of Hypertension & Vascular Risk Unit. Nephrology Department, Parc de Salut Mar
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ATHAN
Record Dates: First submitted 2020-03-04; First posted 2020-07-09 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Treatment Adherence
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Interventional, prospective, randomized, controlled, parallel groups, open study
Who Masked: Participant
Masking Description: Patients are not knowledged whether they are allocated to the control group or to the interventional group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): usual medical follow-up
- Intervention (Active Comparator): Implementation of a specific program to improve therapeutic adherence
  Interventions: Other: implementation of a specific program to improve therapeutic adherence

INTERVENTIONS:
Other: implementation of a specific program to improve therapeutic adherence — 1. Discussion of risks associated with high BP;aims,healthy lifestyle options.
  2. Individualized educational intervention:verbal, written,audiovisual information. Evaluation of knowledge of prescribed drugs.
  3. Behavioral counseling.training patients to participate in their own care, while positively modifying their skills or routines (i.e. pill boxes,calendars,specific measures to remind the patient taking drugs,adapt the regimen to atient's daily routine).
  4. Socio-psycho-affective interventions.
  5. Reminder systems: phone,email,alarm on the mobile phone.
  6. Simplification as far as possible of therapeutic scheme.
  7. Explanation of prescribed medications (name&dosage), correct intake.
  8. Explanation of possible side effects and what to do if they happen. Facilitate a contact.
  9. Advise and training on home blood pressure self-measurement.
  10. Verbal, written and/or audiovisual information and the online patients'section of scientific societies addresses will be provided.
  Arms: Intervention

SUMMARY:
In hypertension, highly prevalent, up to 10-15% of hypertensive patients have uncontrolled blood pressure despite being treated with ≥3 drugs, which is known as resistant hypertension. Resistant arterial hypertension, together with difficult-to-control hypertension, has a worse cardiovascular prognosis than controlled hypertension. In addition, data on therapeutic adherence in arterial hypertension show that 1 in 2 hypertensive patients do not fully or partially comply with the indicated therapeutic prescription. The determination of antihypertensive drugs or their metabolites in urine seems to be a good indicator of therapeutic adherence. On the other hand, the implementation of a specific program to improve knowledge of the disease and its risks and promote therapeutic adherence could improve the control of hypertension and reduce the associated morbidity and mortality.

DETAILED DESCRIPTION:
Objective: To assess whether the implementation of a specific action plan to improve adherence for 3 months results in reduced peripheral 24h-systolic blood pressure (SBP) in patients with resistant hypertension (RH) or uncontrolled hypertension with 2 antihypertensive drugs.

Method: interventional, prospective, randomized, controlled, parallel groups, open study of a cohort of 150 consecutively recruited patients with RH (office SBP ≥140mmHg and/or diastolic blood pressure ≥90mmHg despite treatment with ≥3 drugs at appropriate doses, one diuretic) or patients with uncontrolled hypertension with 2 antihypertensive drugs, with ambulatory 24h-BP ≥130 and / or 80mmHg. The partially or completely non-adherent patients (confirmed by determination of antihypertensive drugs in urine) will be randomized (1: 1) to receive a specific program to improve adherence (intervention group) or routine follow-up (control group), with office BP measurement and determination of antihypertensive drugs in urine at pre-randomization, 3, 6 and 12 months; peripheral and central 24h-ambulatory BP monitoring will be performed at pre-randomization, at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* patients aged ≥18 years
* diagnosis of resistant hypertension with treatment superior to 3 drugs at maximum dose, one of them being a diuretic
* uncontrolled hypertension treated with 2 drugs at the maximum effective doses tolerated
* the prescribed treatment must be stable for the last 2 months
* given informed consent

Exclusion Criteria:

* secondary arterial hypertension
* pregnant women
* Impossibility to perform a 24-hour blood pressure monitoring, or poor quality results.
* Recent history of major vascular episode
* patients receiving treatment with Barnidipino / Felodipine / Lercanidipine / Manidipine / Nifedipine / Verapamil / Eplerenone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in 24h-systolic blood pressure. | 3 months
  Comparison between groups of change in 24-hour-systolic blood pressure provided by 24h-ambulatory blood pressure monitoring 3 months after randomization

SECONDARY OUTCOMES:
Variation in the degree of therapeutic compliance | 3 months
  Comparison between groups of therapeutic compliance variation according to the determination of drugs or their metabolites in urine, i.e., percentage of non-adherent patients that become fully antihypertensive treatment adherent after the implementation of the specific program to improve therapeutic adherence, as compared to the same percentage of the group who do not receive this specific program

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital del Mar, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No